CLINICAL TRIAL: NCT02843399
Title: Clinical and Economic Outcomes of Patients With Type 2 Diabetes Mellitus Initiating Bydureon and Glargine
Brief Title: Economic Outcomes of EQW (Exenatide Once Weekly) vs. IG (Insulin Glargine) in T2D Patients Who Are New to Injectable Therapy
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: Truven health (Unknown)
Responsible Party: Sponsor
Other Study IDs: D5551R00012
Record Dates: First submitted 2016-07-21; First posted 2016-07-25 (Estimated); Last update posted 2017-12-15 (Actual); Status verified 2017-12

CONDITIONS: Diabetes Mellitus Type 2
Keywords: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Exenatide once weekly (EQW): EQW cohort includes patients with one or more outpatient prescription claims for EQW between 2012 and 2015.
- Insulin Glargine (IG): IG cohort includes patients with one or more outpatient prescription claims for IG between 2012 and 2015

SUMMARY:
Primary objective of this study is to compare diabetes-related healthcare utilization and costs in patients initiating exenatide once weekly vs insulin glargine.

DETAILED DESCRIPTION:
This retrospective, observational cohort analysis will assess medical and pharmacy claims for adult patients with type 2 diabetes from the Truven Health MarketScan® Commercial and Medicare Supplemental claims databases between 2011 and 2015. Diabetes-related healthcare utilization and costs will be measured as a primary outcome. Secondary outcomes include all-cause healthcare utilization and costs, major adverse cardiovascular event (MACE)-related utilization and costs, and medically attended hypoglycemia events.

ELIGIBILITY:
Inclusion Criteria:

1. One or more outpatient prescription claim for EQW (Exenatide Once Weekly) vs. IG (Insulin Glargine) between February 1, 2012, and June 30, 2014 (date of first claim = index date; medication to which first claim corresponds = index therapy).
2. Aged 18 or older as of the index date.
3. Continuous enrollment in medical and pharmacy benefits for 12 months before (baseline period) and 12 months after (follow-up period) the index date. (6 months follow-up will be provided to determine the effect on sample size.)
4. One or more medical claims with a diagnosis code for T2DM (ICD-9-CM 250.x0 or 250.x2) in the baseline period or on the index date.

Exclusion Criteria:

1. No outpatient prescription claims for any injectable glucose-lowering medication during the baseline period (GLP-1RA or insulins).
2. No medical claims with a diagnosis (or procedure, where appropriate) code indicative for type 1 diabetes mellitus (ICD-9-CM 250.x1 or 250.x3), gestational diabetes (ICD-9-CM 648.8x), or pregnancy or childbirth in the baseline or follow-up periods.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Commercial Insurance
Sampling Method: Non-Probability Sample
Enrollment: 15498 (Actual)
Dates: Start 2016-08-15 (Actual); Primary Completion 2016-12-15 (Actual); Study Completion 2016-12-15 (Actual)

PRIMARY OUTCOMES:
Diabetes-related HCRU/costs | Up to 12 months
  Compare diabetes-related healthcare utilization and costs in patients initiating EQW (Exenatide Once Weekly) vs. IG (Insulin Glargine)

SECONDARY OUTCOMES:
Overall HCRU/Costs | Up to 12 Months
  To compare overall healthcare utilization and costs in patients initiating EQW (Exenatide Once Weekly) vs. IG (Insulin Glargine)
MACE-related HCRU/Costs | Up to 12 Months
  To compare major adverse cardiovascular event (MACE)-related healthcare utilization and costs in patients initiating EQW (Exenatide Once Weekly) vs. IG (Insulin Glargine)
Medical Hypoglycemic events | Up to 12 Months
  To compare rates and costs of medically attended hypoglycemia in patients initiating EQW (Exenatide Once Weekly) vs. IG (Insulin Glargine)

OTHER OUTCOMES:
Composite of A1C <7%/no weight gain/no hypoglycemia | Up to 12 Months
  The exploratory objective of this analysis is to compare attainment of a composite endpoint, and attainment of each of the individual components thereof separately, comprising an HbA1c less than 7%, no weight gain, and no hypoglycemia in patients initiating EQW (Exenatide Once Weekly) vs. IG (Insulin Glargine). This will be conducted among a subset of patients with available laboratory data.

CONTACTS AND LOCATIONS:
Overall Officials: Eric T. Wittbrodt, PharmD, MPH, Study Director — AstraZeneca
Locations (1):
- Research site, Wilmington, Delaware, United States

REFERENCES:
- See also: Synopsis_D5551R00012 — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4406&filename=Synopsis_D5551R00012.pdf